CLINICAL TRIAL: NCT04953494
Title: Pleiotropy and Mechanism of Peripheral Nerve Related Genes in the Progression of Amyotrophic Lateral Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021051
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amyotrophic lateral sclerosis patients group
  Interventions: Diagnostic Test: Patient information collection, exon sequencing and follow-up.

INTERVENTIONS:
Diagnostic Test: Patient information collection, exon sequencing and follow-up. — Clinical baseline data, disease characteristics, auxiliary examination results, EMG examination results, drug use and other information were collected. 4-6ml peripheral blood was collected for exon sequencing. The patients were followed up every three months by a specialist in the form of outpatient or telephone.

SUMMARY:
This study will establish a comprehensive exon database of ALS patients, lay the foundation for screening the genes related to the occurrence and development of the disease, support the theory of ALS disease progression from peripheral to central, and reveal the correlation between the functional level of peripheral nerve and the prognosis of the disease at the gene level for the first time, and provide the basis for the mechanism research at the molecular level.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease that selectively invades superior and inferior motor neurons. Because there is no effective treatment, it is urgent to find the risk factors of ALS to guide the prevention and slow down the disease progression. In the early stage of the disease, the peripheral motor injury is more rapid and sensitive than the central response, which is an ideal window to observe the state of the disease. Protecting peripheral nerve integrity and maintaining its function can slow down the death of superior neurons, effectively relieve symptoms and prolong survival time, which has also been confirmed in patients with multiple stem cell-derived motor neurons and SOD1 G93A disease model mice. Reexamination of the role of peripheral motor nerve related factors in the development of ALS is of great significance for the study of disease mechanism, clinical classification, prognosis, evaluation of drug trial efficacy and individualized treatment plan. Previous studies have shown that NEFL gene, as the coding gene of light chain of neuron cytoskeleton, is closely related to axonal function, and its polymorphism is related to the occurrence and severity of axonal Charcot Marie Tooth disease. Exploring the role of similar peripheral nerve related genes in the progression of ALS will help us better understand the disease from the genetic level, establish an accurate and stable prognosis prediction model, and guide early treatment. This study will establish a comprehensive exon database of ALS patients, lay the foundation for screening the genes related to the occurrence and development of the disease, support the theory of ALS disease progression from peripheral to central, and reveal the correlation between the functional level of peripheral nerve and the prognosis of the disease at the gene level for the first time, and provide the basis for the mechanism research at the molecular level.

ELIGIBILITY:
Inclusion Criteria:

1. Since February 2021, he has been in the Department of Neurology, the Third Hospital of Beijing Medical University. He was diagnosed amyotrophic lateral sclerosis according to the revised EI Escorial diagnostic criteria of 2004 edition, and the patients within one year of onset.
2. Informed consent has been signed.

Exclusion Criteria:

1. Patients with ALS like syndrome caused by autoimmune diseases, paraneoplastic syndrome and simple demyelinating lesions were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Amyotrophic lateral sclerosis patients in Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
death | until the patient dies, usually 1-10 years after diagnosis.
  patients' death
invasive breathing | until the patient has invasive breathing, usually 1-10 years after diagnosis.
  The patient uses a ventilator to maintain breathing

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No